CLINICAL TRIAL: NCT06744738
Title: Pharmacist-led Intervention on Hemodialysis Patients' Therapy Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thuraya Safaa Ibrahim (Other)
Responsible Party: Sponsor-Investigator, Thuraya Safaa Ibrahim, Principal Investigator, University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RECAUCP8720246
Record Dates: First submitted 2024-12-16; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Hemodialysis; End Stage Renal Disease Requiring Hemodialysis
Keywords: Adherences; Chronic kidney disease; ESRD; Behavioral intervention
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care (No Intervention): The usual care group received the usual care offered by the center to all patients, which included printed, paper-based, and verbal instructions. The written material included knowledge about diet recommendations for dialysis patients based on National Kidney Foundation recommendations. Verbal instructions were provided by the physician, including information regarding their medications, dialysis, diet, and fluid intake based on their condition and monthly lab results. Medications are provided to all patients at no cost, and pharmacists provide instructions on how to use them.
- pharmacist-led behavioral change technique (Experimental): The intervention was developed based on the behavior change technique taxonomy (v1). This intervention was designed to improve adherence to all therapeutic aspects of hemodialysis patients, including the dialysis program, medications, diet, and fluids. Additionally, the effect of the pharmacist intervention on physiological indices (serum potassium, total calcium, phosphate, IDWG, and hemoglobin) was examined.
  The program was explicitly created for implementation in an actual setting, ensuring that the time allocation for participants and facilitators (the party responsible for conducting the PL-BCT) remained reasonable in most contexts.
  The BCT components were developed after the identification and coding of the BCTs from previous interventional studies that contain behavioral components and result in positive effects on one or more hemodialysis patients' adherence domains toward their therapeutic regimen (dialysis program, medications, diet, and fluid).
  Interventions: Behavioral: Pharmacist led behavioral change technique

INTERVENTIONS:
Behavioral: Pharmacist led behavioral change technique — The intervention was developed based on the behavior change technique taxonomy (v1). This intervention was designed to improve adherence to all therapeutic aspects of hemodialysis patients, including the dialysis program, medications, diet, and fluids. Additionally, the effect of the pharmacist intervention on physiological indices (serum potassium, total calcium, phosphate, IDWG, and hemoglobin) was examined.
  The program was explicitly created for implementation in an actual setting, ensuring that the time allocation for participants and facilitators (the party responsible for conducting the PL-BCT) remained reasonable in most contexts.
  The BCT components were developed after the identification and coding of the BCTs from previous interventional studies that contain behavioral components and result in positive effects on one or more hemodialysis patients' adherence domains toward their therapeutic regimen (dialysis program, medications, diet, and fluid).
  Arms: pharmacist-led behavioral change technique

SUMMARY:
A parallel-group, cluster-randomized, controlled trial designed to evaluate if hemodialysis patients benefit from BCT. The study includes two groups: usual care and pharmacist-led intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years of age), chronic kidney disease patients on standard in-center hemodialysis for at least three months, patients receiving 4 hours per session, moderate to poor adherence to their therapeutic regimen according to End Stage Renal Disease Adherence Questionnaire (ESRD-AQ) at the time of inclusion

Exclusion Criteria:

* Switching from hemodialysis to peritoneal dialysis, receiving transplantation during the research period, inability to communicate for any reason (cognitive impairment, hearing and visual loss, etc.), hemodialysis patients with viral hepatitis, and patient refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
End Stage Renal Disease Adherence Questionnaire (ESRD-AQ) scores | At the start of the study, and after one month of the start of the study.
  The ESRD-AQ is a comprehensive tool that records critical elements of patients' treatment history: self-reported treatment adherence (including HD attendance, prescriptions, fluid restrictions, and dietary recommendations); perceptions regarding adherence behaviors; and justifications for nonadherence. ESRD-AQ consists of 46 questions, scores range from 0 to 1,200, with higher scores signify better adherence. Scores are divided into three ranges to identify adherence behavior (good adherence scores range between 1000 to 1200, moderate adherence scores range between 700 to 999, and poor adherence scores are less than 700). The scores were distributed over the four dimensions as follows: adherence to HD sessions (scores 0 - 600), adherence to dietary recommendations (scores 0 - 200), adherence to medications (scores 0 - 200), and adherence to fluid restriction (scores 0 - 200)

SECONDARY OUTCOMES:
Serum Phosphate | At the start of the study, and after one month of the start of the study.
  Serum Phosphate levels measurement
Interdialytic weight gain (IDWG) | At the start of the study, and after one month of the start of the study.
  Interdialytic weight gain (IDWG) Assessment
Total serum Calcium | At the start of the study, and after one month of the start of the study.
  Total serum Calcium measurement
Hemoglobin levels | At the start of the study, and after one month of the start of the study.
  Measurement of patients Hemoglobin levels

CONTACTS AND LOCATIONS:
Locations (1):
- Baghdad Medical City, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ansaf TS, Al-Hamadani FY, Brown S, James DH. Pharmacist-led behavioral change intervention improves adherence and clinical outcomes among hemodialysis patients. Sci Rep. 2025 Sep 29;15(1):33661. doi: 10.1038/s41598-025-18082-y. PMID 41023004